CLINICAL TRIAL: NCT06550999
Title: Patient Satisfaction and Cosmetic Outcomes in Adhesive Strip Versus Suture Repair for Simple Facial Lacerations: A Randomized Controlled Trial
Brief Title: Patient Satisfaction and Cosmetic Outcomes in Adhesive Strip Versus Suture Repair for Simple Facial Lacerations
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Irvine (Other)
Responsible Party: Principal Investigator, Jeffry Nahmias, MD, Health Sciences Professor, University of California, Irvine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 4338
Record Dates: First submitted 2024-07-11; First posted 2024-08-13 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Facial Laceration
Keywords: Adhesive strips; Sutures; Laceration repair; Cosmesis; Scar healing
MeSH Terms: interventions — Sutures

STUDY DESIGN:
Intervention Model Description: This is a prospective, single-blinded, randomized controlled trial taking place in a single center. Patients will be identified in the emergency room as they present to the hospital and meet eligibility criteria. Following informed consent, patients will be randomized in a 1:1 ratio to either the adhesive strip repair or the suture repair group. Randomization will be dictated by a validated online software utilizing the Wichmann-Hill random number generator. Randomization and allocation concealment will be managed by a nominated independent individual(s) not involved in patient care or data extraction/analysis. A password-protected randomization database that is only accessible to the study team will be utilized.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Following informed consent, patients will be randomized to either the adhesive strip repair group or the suture repair group for their facial laceration. The patient and care provider will therefore know which group they are part of. Randomization and allocation concealment will be managed by a nominated independent individual(s) not involved in patient care or data extraction/analysis. A password-protected randomization database that is only accessible to the study team will be utilized. The investigator and outcomes assessor will be blinded to the group assignments.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Adhesive strip repair (Experimental): In this arm, patients will have their facial laceration properly cleaned and repaired with adhesive strips.
  Interventions: Device: Laceration repair with adhesive strips
- Suture repair (Experimental): In this arm, patients will have their facial laceration properly cleaned and repaired with sutures of any material.
  Interventions: Procedure: Laceration repair with sutures

INTERVENTIONS:
Device: Laceration repair with adhesive strips — Repair of the patient's facial laceration with adhesive strips
  Other Names: Adhesive strips; Steri-Strips; STERI-STRIP ANTIMICROBIAL SKIN CLOS
  Arms: Adhesive strip repair
Procedure: Laceration repair with sutures — Repair of the patient's facial laceration with sutures
  Arms: Suture repair

SUMMARY:
There are a variety of techniques utilized to close lacerations, including but not limited to, traditional sutures, staples, adhesive strips, and skin glue. While closing open wounds and preventing infection are the primary goals of laceration repair, physicians are also concerned with minimizing scar formation and providing the best cosmetic outcomes for the patient. Specifically, the skin on the face is a sensitive area where cosmetic outcome is of high importance, and several laceration repair techniques have been devised for closing facial wounds.

Sutures have traditionally been used to close wounds in various types of tissue, and it is still very commonly used in the clinical setting. Adhesive strips (also known under the brand names of Steri-Strips, Curi-strips, Nichi-Strips, and Suture Strips) are another method to repair lacerations superficially. Due to their superficial application and ease of use, adhesive strips may help minimize scar formation and may result in less pain and complications for the patient when compared to conventional sutures.

Therefore, the aim of this study is to determine whether repair of small, simple facial lacerations with adhesive strips results in better patient experiences and better cosmetic outcomes than sutures. The investigators hypothesize that wounds repaired with adhesive strip will have higher patient satisfaction scores and better cosmetic outcomes.

DETAILED DESCRIPTION:
This is a prospective, single-blinded, randomized controlled trial taking place in a single center. Patients will be identified in the emergency room as they present to the hospital and meet eligibility criteria. Following informed consent, patients will be randomized in a 1:1 ratio to either the adhesive strip repair or the suture repair group. Randomization will be dictated by a validated online software utilizing the Wichmann-Hill random number generator. A password-protected randomization database that is only accessible to the study team will be utilized.

After randomization to their respective laceration repair group, patients will be surveyed by the study team to assess their experience, satisfaction, and pain scores during the laceration repair. Approximately two months after their initial laceration repair, the patients will be contacted securely via phone call or email to assess if they had any complications and to assess their satisfaction and cosmetic rating of their laceration scar. Additionally, the subjects will be instructed to take pictures and/or videos of their scar and send it securely to the study team via UCI Epic MyChart (or a HIPAA-compliant encrypted email if MyChart is unavailable). These photos and videos will be de-identified and stored securely on a password-encrypted folder where a blinded evaluator will score the scars with a validated scar assessment tool. Patients will be instructed to only take photos/videos of their scar area and not any other major areas of their face that can be identified. Following the conclusion of the study, all patient identifiers and photos/videos will be destroyed to preserve patient privacy.

All survey data will be collected and entered into a REDCap database. Data collection will include demographics, phone/email contact information, patient satisfaction scores with the laceration repair, patient pain scores, patient scar cosmetic rating, presence of complications, and patient responses to questions about their general experience during the laceration repair and healing time period.

ELIGIBILITY:
Inclusion Criteria:

* All adult (>18-years-old)
* Small (<2.5 cm) and simple facial lacerations requiring repair

Exclusion Criteria:

* Patients less than 18 years old
* Pregnant females
* Incarcerated individuals

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2026-08 (Estimated); Primary Completion 2028-05 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Patient pain score | Assessed immediately after the intervention
  Visual analogue scale (VAS) - 10-cm line representing a continuum from "no pain" to "worst pain imaginable"
Patient's satisfaction and experience during laceration repair | Assessed immediately after the intervention
  Measured on a Likert-scale (very dissatisfied, dissatisfied, neutral, satisfied, very satisfied) and measured with a visual analogue scale (VAS) ("not satisfied" and to "fully satisfied")
Patient's cosmetic score of the laceration immediately after repair | Assessed immediately after the intervention
  Measured on a visual analogue scale (VAS) - 100-mm visual analogue scale for cosmetic assessment of wound (0 = worst scar and 100 = best scar)
Patient's cosmetic score of the laceration scar | Assessed two months after the intervention
  Measured via the Patient and Observer Scar Assessment Scale (POSAS) - a validated cosmetic score assessment for wounds from the patient's perspective. Each item of the POSAS is rated on a 5-point score. The lowest score is '1', which corresponds to the situation of normal skin (i.e. normal pigmentation, no itching). Score 5 equals the largest difference from normal skin (i.e. the worst imaginable scar or sensation).
Evaluator's cosmetic score of the wound assessed from a photograph | Assessed two months after the intervention
  Measured on the Stoney Brook Scar Evaluation Scale (SBSES) - a validated cosmetic score assessment of scars from the observer's perspective using a photograph. Scars are assigned either 0 or 1 point each for the presence or absence of the following: width greater than 2 mm, elevation or depression, discoloration, suture or staple marks, and overall poor appearance. A total cosmetic score is generated by adding the individual scores from each category ranging from 0 (worst) to 5 (best)

SECONDARY OUTCOMES:
Time to repair laceration | Assessed immediately after the intervention
  The amount of time lapsed in repairing the laceration
Laceration/scar length and width | Assessed immediately after the intervention and two months after the intervention
  The length and width in centimeters of the subject's laceration/scar
Complications during and/or after the repair | Assessed immediately after the intervention and two months after the intervention
  Complications during the procedure will be evaluated by the study team by retrieving data from the medical chart, observing the laceration repair in real time, or surveying the patient after the laceration repair. Post-procedural complications will be evaluated by following up with patients via phone call or secure email

CONTACTS AND LOCATIONS:
Overall Officials: Jeffry Nahmias, M.D., Principal Investigator — University of California, Irvine
Locations (1):
- University of California Irvine, Orange, California, United States

IPD SHARING:
Plan to Share IPD: No
No plan to share IPD